CLINICAL TRIAL: NCT04790253
Title: PRophylactic Cerebral Irradiation or Active MAgnetic Resonance Imaging Surveillance in Small-cell Lung Cancer Patients (PRIMALung Study)
Acronym: PRIMALung
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Collaborators: UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EORTC-1901-LCG
Record Dates: First submitted 2021-03-05; First posted 2021-03-10 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Limited Stage Small Cell Lung Cancer; Extensive-stage Small-cell Lung Cancer
Keywords: Prophylactic cerebral Irradiation; small cell lung cancer; PCI
MeSH Terms: conditions — Small Cell Lung Carcinoma

STUDY DESIGN:
Intervention Model Description: After eligibility checks, patients will be randomized between the 2 arms, and stratified by stage of disease (limited versus extensive), immunotherapy as part of the first-line treatment (yes/no), and ECOG Performance Status (0 or 1 versus 2).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PCI followed by brain MR surveillance (Active Comparator): Prophylactic cranial irradiation will be delivered at the dose of 25 Gy in 10 fractions to the whole brain.
  Patients must have a brain MRI performed within 28 days before randomisation and at 3, 6, 9, 12, 18 and 24 months.
  Extracranial imaging is recommended and will be performed per institutional standards at the discretion of the treating physician.
  Interventions: Radiation: Prophylactic cranial irradiation
- MRI Active Surveillance (No Intervention): Patients must have a brain MRI performed within 28 days before randomisation and at 3, 6, 9, 12, 18 and 24 month. Clinical evaluation will be performed every 3 months.

INTERVENTIONS:
Radiation: Prophylactic cranial irradiation — Prophylactic cranial irradiation (PCI) is a technique used to combat the occurrence of metastasis to the brain in highly aggressive cancers that commonly metastasize to brain, most notably small-cell lung cancer.
  Arms: PCI followed by brain MR surveillance

SUMMARY:
In this phase III study, the primary objective is to test with a one-sided significance of 5% whether for the treatment of small cell lung cancer (SCLC) patients, brain MRI surveillance alone is non-inferior in terms of overall survival compared to prophylactic cranial irradiation (PCI) combined with brain MRI surveillance in the entire study population.

DETAILED DESCRIPTION:
The primary objective is to test with a one-sided significance of 5% whether for the treatment of small cell lung cancer (SCLC) patients, brain MRI surveillance alone is non-inferior in terms of overall survival compared to prophylactic cranial irradiation (PCI) combined with brain MRI surveillance in the entire study population under the treatment policy strategy.

The secondary objectives are:

* To test with a one-sided type I error of 2.5% whether brain MRI surveillance is superior in terms of cognitive failure free survival (CFFS) compared to prophylactic cranial irradiation (PCI) combined with brain MRI surveillance in the study population.
* To test with a one-sided type I error of 2.5% whether brain MRI surveillance is superior in terms of global health status/QoL and cognitive functioning according to EORTC QLQ-C30 questionnaire compared to prophylactic cranial irradiation (PCI) combined with brain MRI surveillance in the study population.
* To evaluate the frequency and severity of toxicities according to CTCAE v5.0 in the two arms in the treated population (i.e. patients who have started treatment).

The exploratory objectives are:

* To compare OS and CFFS between the arms within the subgroups of patients with LS and ES disease.
* To compare OS and CFFS between the arms within the subgroups: HA-PCI or not, first-line immunotherapy or not, memantine or not.
* To compare cognitive failure free survival (CFFS) rate at 12 months after randomization between the arms.
* To compare the cumulative incidence of cognitive failures with death as a competing risk between the arms.
* To compare brain-metastasis-free survival (BMFS) between the arms.
* To compare progression free survival (PFS) between the arms.
* To compare time to brain-metastasis-attributed death (TBMAD) between the arms.
* To compare other QoL scales according to EORTC QLQ-C30 and QLQ-BN20 questionnaires between arms.
* To evaluate the cost-effectiveness of MRI surveillance alone versus MRI surveillance combined with PCI.
* To collect blood for biobanking.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Histologically/cytologically proven diagnosis of SCLC
* Limited and extensive stage
* LS SCLC: Stage I-III (T any, N any, M0, according to UICC TNM staging v8.0) that can be safely treated with definitive radiation doses. Excludes T3-4 due to multiple lung nodules that are too extensive or have tumour/nodal volume that is too large to be encompassed in a tolerable radiation plan.
* ES SCLC: Stage IV (T any, N any, M 1a/b), or T3-4 due to multiple lung nodules that are too extensive or have tumour/nodal volume that is too large to be encompassed in a tolerable radiation plan.
* Completed standard therapy prior to randomization:
* For patients with LS-SCLC, this includes a combination of 4-6 cycles of platinum-based doublet chemotherapy and either definitive thoracic radiotherapy (including SBRT for early-stage T1-2 N0 M0 disease who do not undergo surgery) or definitive surgical resection; thoracic radiation in addition to definitive surgical resection is allowed at the discretion of the treating physician, but is not mandated.
* For patients with ES-SCLC, this includes 4-6 cycles of platinum-based doublet chemotherapy either with or without thoracic radiotherapy

  o Immunotherapy concurrent with and/or adjuvant to standard therapy is allowed at the discretion of the treating physician.
* Absence of progressive disease after completed standard therapy on systemic imaging (computed tomography (CT) or magnetic resonance imaging (MRI) of Chest/Abdomen/Pelvis and brain MRI), 28 days before randomization.
* Absence of brain metastases or leptomeningeal disease after completed standard therapy on systemic imaging (computed tomography (CT) or magnetic resonance imaging (MRI) of Chest/Abdomen/Pelvis and brain MRI), within 28 days before randomization.
* Interval from day 1 of last cycle of chemotherapy to randomization of ≤8 weeks
* ECOG PS ≤ 2
* Estimated creatinine clearance ≥ 30 mL/min as calculated using the MDRD formula
* Women of child bearing potential (WOCBP) must have a negative serum pregnancy test within 3 days prior to randomization.

Note: women of childbearing potential are defined as premenopausal females capable of becoming pregnant (i.e. females who have had any evidence of menses in the past 12 months, with the exception of those who had prior hysterectomy). However, women who have been amenorrheic for 12 or more months are still considered to be of childbearing potential if the amenorrhea is possibly due to prior chemotherapy, antioestrogens, low body weight, ovarian suppression or other reasons.

* Patients Women of childbearing / reproductive potential should use adequate birth control measures, as defined by the investigator, during the entire period of the radiotherapy treatment study participation and for at least 30 days after the last dose of radiotherapy. A highly effective method of birth control is defined as a method which results in a low failure rate (i.e. less than 1% per year) when used consistently and correctly. Such methods include:
* Combined (oestrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal)
* Progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable)
* Intrauterine device (IUD)
* Intrauterine hormone-releasing system (IUS)
* Bilateral tubal occlusion
* Vasectomized partner
* Sexual abstinence (the reliability of sexual abstinence needs to be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient)
* Female subjects who are breast feeding should discontinue nursing prior to the first dose of radiotherapy and during the entire period of the radiotherapy treatmentuntil 30 days after the administration of the last dose of radiotherapy.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
* Before patient registration/randomization, written informed consent must be given according to ICH/GCP, and national/local regulations.

Exclusion Criteria:

* Prior radiotherapy to the brain or whole brain radiotherapy. Note: Patients who have undergone prior stereotactic radiosurgery for benign tumours or conditions (e.g., acoustic neuroma, grade I meningioma, trigeminal neuralgia) may be considered on a case-by-case basis. Discussion with EORTC Headquarters is mandatory, before the randomization.
* Known contraindication to imaging tracer or any product of contrast media, such as allergy or insufficient renal function. Known contraindication to MRI, such as implanted metal devices or foreign bodies.
* Other active hematologic or solid tumour malignancy requiring current active treatment.
* Any unresolved toxicities from prior therapy (e.g., chemotherapy, radiotherapy) greater than CTCAE grade 2 (according to CTCAE v5.0) at the time of randomization.
* Patient with severe active comorbidities, defined as follows:
* Unstable angina and/or congestive heart failure requiring hospitalization within 6 months prior to randomization
* Transmural myocardial infarction within 6 months prior to randomization
* Acute infection requiring treatment at the time of randomization
* Chronic obstructive pulmonary disease exacerbation or other acute respiratory illness precluding study therapy at the time of randomization
* Severe hepatic disease defined as a diagnosis of Child-Pugh class B or C hepatic disease
* HIV positive with CD4 count < 200 cells/microliter. Note: patients who are HIV positive are eligible, provided they are under treatment with highly active antiretroviral therapy (HAART) and have a CD4 count ≥ 200 cells/microliter within 16 weeks prior to randomization.
* Any severe comorbidity that in the opinion of the Investigator might hamper the participation to the study and/or the treatment administration.
* Severe neurological (including dementia and epilepsy) or psychiatric disorder requiring active treatment.
* Any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before randomization in the trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2022-10-27 (Actual); Primary Completion 2028-04 (Estimated); Study Completion 2028-04 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 12 Months
  The primary objective is to test with a one-sided significance of 5% whether for the treatment of small cell lung cancer (SCLC) patients, brain MRI surveillance alone is non-inferior in terms of overall survival compared to prophylactic cranial irradiation (PCI) combined with brain MRI surveillance in the entire study population

SECONDARY OUTCOMES:
cognitive failure free survival | 12 Months
  To test with a one-sided type I error of 2.5% whether brain MRI surveillance is superior in terms of cognitive failure free survival (CFFS) compared to prophylactic cranial irradiation (PCI)
Quality of Life | 12 Months
  To show that brain MRI surveillance is superior in terms of global health status/QoL and cognitive functioning according to EORTC QLQ-C30 questionnaire compared to prophylactic cranial irradiation (PCI) combined with brain MRI surveillance
Safety profiling | 12 Months
  To evaluate the frequency and severity of toxicities according to CTCAE v5.0 in the two arms in the treated population (i.e. patients who have started treatment).

CONTACTS AND LOCATIONS:
Overall Officials: Corinne Faivre-Finn, MD, Principal Investigator — The Christie NHS Foundation Trust; Antonin Levy, MD, Principal Investigator — Centre Gustave Roussy
Locations (41):
- Medical University of Graz - Radio-oncology, Graz, Austria
- Belgium (5):
  - Institut Jules Bordet, Anderlecht
  - Universitair Ziekenhuis Antwerpen, Edegem
  - AZ Groeninge Kortrijk - Campus Kennedylaan, Kortrijk
  - C.H.U. Sart-Tilman, Liège
  - Gasthuiszusters van Antwerpen - GasthuisZusters Antwerpen - Sint-Augustinus, Wilrijk
- France (13):
  - Institut Sainte Catherine (UNICANCER), Avignon
  - Centre D'Onco. & Radioth. De Haute Energie Du Pays Basque (UNICANCER), Bayonne
  - Institut Bergonie (UNICANCER), Bordeaux
  - Centre Francois Baclesse (CLCC) (UNICANCER), Caen
  - CHU de Dijon - Centre Georges-Francois-Leclerc (UNICANCER), Dijon
  - Centre Hospitalier Departemental Vendee (UNICANCER), La Roche-sur-Yon
  - Institut Paoli-Calmettes (UNICANCER), Marseille
  - Institut du Cancer de Montpellier (UNICANCER), Montpellier
  - Centre Catalan d'Oncologie (UNICANCER), Perpignan
  - CHU de Lyon - Hopital Lyon Sud (UNICANCER), Pierre-Bénite
  - Centre Henri Becquerel (UNICANCER), Rouen
  - Institut de Cancerologie Strasbourg Europe (UNICANCER), Strasbourg
  - Gustave Roussy (UNICANCER), Villejuif
- Universitaetsklinikum Aachen AOR - Medizinische Fakultaet der RWTH, Aachen, Germany
- Italy (5):
  - IRCCS Azienda Ospedaliera Universitaria San Martino "IST" - IRCCS - AUO San Martino - IST, Genova
  - ULSS 9 Scaligera Veneto - Azienda Unita Locale Socio-Sanitaria N. 9-Mater Salutis Hospital, Legnago
  - Fondazione IRCCS - Policlinico San Matteo, Pavia
  - ASST-Bergamo Ospedale Treviglio-Caravaggio, Treviglio
  - Azienda Ospedaliera Universitaria Integrata Verona - Ospedale Borgo Roma, Verona
- Poland (2):
  - Medical University Of Gdansk, Gdansk
  - Regional Cancer Centre, Olsztyn
- Spain (3):
  - Hospital Universitario Badajoz, Badajoz
  - Hospital Insular De Gran Canaria, Las Palmas de Gran Canaria
  - Hospital Universitario Puerta De Hierro, Majadahonda
- Switzerland (4):
  - Inselspital, Bern
  - Reseau Hospitalier Neuchatelois - RHNe - La Chaux de Fonds, La Chaux-de-Fonds
  - Kantonsspital St Gallen, Sankt Gallen
  - UniversitaetsSpital Zurich, Zurich
- United Kingdom (7):
  - University Hospitals Bristol NHS Foundation Trust - Bristol Haematology And Oncology Centre, Bristol
  - NHS Lothian - Western General Hospital, Edinburgh
  - Maidstone & Tunbridge Wells NHS Trust - Maidstone Hospital, Maidstone
  - The Christie NHS Foundation Trust, Manchester
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - Sheffield Teaching Hospitals NHS Foundation Trust - Weston Park Hospital, Sheffield
  - Royal Marsden Hospital - Sutton, Sutton